CLINICAL TRIAL: NCT03002974
Title: A Randomized, Double-blind, Active-control, Multicenter, Efficacy and Safety Study of 2 Dose Levels of Subcutaneous Anakinra Compared to Intramuscular Triamcinolone in the Treatment of Acute Gouty Arthritis, Followed by an Extension Period of up to 2 Years
Brief Title: A Study to Evaluate Efficacy and Safety of Anakinra in the Treatment of Acute Gouty Arthritis
Acronym: anaGO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sobi.ANAKIN-401
Record Dates: First submitted 2016-12-13; First posted 2016-12-26 (Estimated); Results first posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-06

CONDITIONS: Acute Gouty Arthritis
Keywords: Gout; Interleukin 1 receptor antagonist; IL-1 receptor antagonist
MeSH Terms: conditions — Gout | interventions — Interleukin 1 Receptor Antagonist Protein; Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Anakinra 100 mg (Experimental): 1 subcutaneous injection of Anakinra 100 mg once daily for 5 days, 1 subcutaneous injection of Placebo to Anakinra 100 mg once daily for 5 days and 1 single intramuscular injection of Placebo to Triamcinolone Acetonide 40 mg
  Interventions: Drug: Anakinra 100 mg; Drug: Placebo to Anakinra 100 mg; Drug: Placebo to Triamcinolone Acetonide 40 mg
- Anakinra 200 mg (Experimental): 2 subcutaneous injections of Anakinra 100 mg (2 syringes) once daily for 5 days and 1 single intramuscular injection of Placebo to Triamcinolone Acetonide 40 mg
  Interventions: Drug: Anakinra 100 mg; Drug: Placebo to Triamcinolone Acetonide 40 mg
- Triamcinolone 40 mg (Active Comparator): 2 subcutaneous injections of Placebo to Anakinra 100 mg once daily for 5 days and 1 single intramuscular injection of Triamcinolone Acetonide 40 mg
  Interventions: Drug: Triamcinolone Acetonide 40 mg; Drug: Placebo to Anakinra 100 mg

INTERVENTIONS:
Drug: Anakinra 100 mg — 100 mg/0.67 mL solution in single-use prefilled syringes for subcutaneous injection
  Other Names: Kineret
  Arms: Anakinra 100 mg; Anakinra 200 mg
Drug: Triamcinolone Acetonide 40 mg — 1 mL intramuscular injection of a 40 mg/mL injectable suspension
  Other Names: Kenalog; Triamcinolone
  Arms: Triamcinolone 40 mg
Drug: Placebo to Anakinra 100 mg — sterile solution for injection (0.67 mL) in a single-use prefilled syringe identical to the anakinra syringe
  Other Names: Placebo Kineret
  Arms: Anakinra 100 mg; Triamcinolone 40 mg
Drug: Placebo to Triamcinolone Acetonide 40 mg — 1 mL intramuscular injectable suspension with identical appearance as the Triamcinolone Acetonide suspension
  Other Names: Placebo Kenalog
  Arms: Anakinra 100 mg; Anakinra 200 mg

SUMMARY:
The purpose of this study is to evaluate how anakinra relieves pain for patients with acute gout that cannot take non-steroidal anti-inflammatory drugs (NSAIDs) and colchicine. The patients will be divided in different treatment groups to compare anakinra to the available drug triamcinolone.

DETAILED DESCRIPTION:
Patients will be randomized to treatment at their first gout flare in the study. The first treatment period will be followed by an extension period during which the patients will receive the same treatment for any subsequent flares within 52 weeks of randomization of last patient in the study. The extension period for the individual patient in the study will be maximum two years (104 weeks). Each new flare treated will initiate a new series of study visits and assessments according to specified schedule of events. Only if a patient experience a new flare after Day 15 of the latest flare they can start a new treatment period. The comparison of primary interest is between anakinra (100 mg and 200 mg combined) and 40 mg triamcinolone, and as a secondary objective the 2 different doses of anakinra will be evaluated as well as assessment for subsequent flares.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed consent
* Patient meeting the American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) 2015 gout classification criteria
* History of ≥1 self-reported flares of gouty arthritis within 12 months
* Current ongoing flare of gouty arthritis characterized by pain intensity
* Currently tender and swollen joint
* Onset of current flare within 4 days
* Intolerant, unresponsive, contraindicated or not appropriate for treatment with NSAIDs and colchicine (both treatment options)
* If on urate-lowering therapy, on a stable dose and regimen
* Women of childbearing potential willing to use adequate contraception

Inclusion criteria for treatment of subsequent flare(s)

* Current flare of gouty arthritis characterized by pain intensity
* Currently tender and swollen joint
* Women of childbearing potential willing to use adequate contraception

Exclusion Criteria:

* Use of specified pain relief medications or biologics (including glucocorticoids, narcotics, paracetamol/acetaminophen, NSAIDs, colchicine, IL-blockers and tumor necrosis factor inhibitors) within specified periods prior to randomization
* Contraindication to triamcinolone
* Polyarticular gouty arthritis involving more than 4 joints
* Rheumatoid arthritis, evidence/suspicion of infectious/septic arthritis, or other acute inflammatory arthritis
* History of malignancy within the past 5 years. Exceptions are basal cell skin cancer, carcinoma-in-situ of the cervix or low-risk prostate cancer after curative therapy.
* Known hypersensitivity to Escherichia coli-derived proteins, Kineret® (anakinra), Kenalog® (triamcinolone acetonide) or any components of the products.
* Known presence or suspicion of active or recurrent bacterial, fungal or viral infections, including tuberculosis, or HIV infection or hepatitis B or C infection
* Presence of severe renal function impairment chronic kidney disease (CKD) stages 4 and 5
* Presence of neutropenia
* Uncontrolled clinically significant hematologic, pulmonary, endocrine, metabolic, gastrointestinal, central nervous system or hepatic disease
* History of myocardial infarction, unstable angina, cerebrovascular events, or coronary artery bypass grafting, New York Heart Association (NYHA) class III or IV heart failure within the previous 3 months
* Patients who have undergone major surgery within 2 weeks, or have an unhealed operation wound/s
* Presence of any medical or psychological condition or laboratory result that in the opinion of the investigator might create risk to the patients or to the study.
* Earlier or current treatment with anakinra
* Pregnant or lactating women
* History of >12 flares overall in the 6 months prior to randomization

Exclusion criteria for treatment of subsequent flare(s):

* Known presence or suspicion of active or recurrent bacterial, fungal or viral infections, including tuberculosis, or HIV infection or hepatitis B or C infection.
* Presence of severe renal function impairment CKD stages 4 and 5
* Presence of neutropenia
* History of myocardial infarction, unstable angina, cerebrovascular events, or coronary artery bypass grafting, NYHA class III or IV heart failure within the previous 3 months
* Patients who have undergone major surgery within 2 weeks or have an unhealed operation wound/s.
* Pregnant or lactating women.
* Presence of any condition or laboratory result that in the opinion of the investigator makes the patient not appropriate for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Ohlman, MD, PhD, Study Director — Swedish Orphan Biovitrum AB
Locations (37):
- United States (37):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Fundamental Research, LLC, Gulf Shores, Alabama
  - Coastal Clinical Research, Inc, Mobile, Alabama
  - Advanced Research Center, Anaheim, California
  - Delta Waves Sleep Disorder and Research Center, Colorado Springs, Colorado
  - Pulmonary Associates of Brandon, Brandon, Florida
  - Meridien Research, Brooksville, Florida
  - Health Awareness, Jupiter, Florida
  - Well Pharma Medical Research, Miami, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Clinical Research Trials of Florida, Tampa, Florida
  - Meridien Research, Inc, Tampa, Florida
  - Kaushik Amin MD, Conyers, Georgia
  - Alta Pharmaceutical Research Center, Dunwoody, Georgia
  - Lemah Creek Clinical Research, Melrose Park, Illinois
  - The Research Group of Lexington, Lexington, Kentucky
  - Clinical Trials Management, Metairie, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Duke University Medical Center, Durham, North Carolina
  - Boiling Springs Medical Research, Inc., Shelby, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Hightop Medical Research Center, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Clinical Research Solutions - Franklin, Franklin, Tennessee
  - Clinical Research Solutions, Smyrna, Tennessee
  - Renaissance Clinical Research and Hypertension Clinic of Texas, PLLC, Dallas, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Accurate Clinical Management, Pasadena, Texas
  - Sun Research Institute, San Antonio, Texas
  - Wade Family Medicine, Bountiful, Utah
  - Ericksen Research & Development, Clinton, Utah
  - Advanced Clinical Research - West Jordan, West Jordan, Utah
  - Commonwealth Clinical Research Specialists, Inc., Richmond, Virginia
  - Corporation Lane Internal Medicine and Research Center, Virginia Beach, Virginia
  - Mileground Physicians, PLLC, Morgantown, West Virginia
  - Clinical Investigations Specialists, Inc., Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saag KG, Khanna PP, Keenan RT, Ohlman S, Osterling Koskinen L, Sparve E, Akerblad AC, Wiken M, So A, Pillinger MH, Terkeltaub R. A Randomized, Phase II Study Evaluating the Efficacy and Safety of Anakinra in the Treatment of Gout Flares. Arthritis Rheumatol. 2021 Aug;73(8):1533-1542. doi: 10.1002/art.41699. Epub 2021 Jul 7. PMID 33605029

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Started | 55 | 56 | 54
Intention To Treat Populatio | 55 | 56 | 54
Safety Population | 54 | 55 | 52
Completed | 35 | 40 | 36
Not Completed | 20 | 16 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg | Total
Number analyzed (Participants) | 55 | 56 | 54 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (10.3) | 53.7 (11.9) | 54.0 (13.1) | 54.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 7 | 22
  Male | 48 | 48 | 47 | 143
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 39 | 38 | 42 | 119
  Race: Black or African American | 15 | 15 | 12 | 42
  Race: Asian | 1 | 3 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 55 | 56 | 54 | 165

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-assessed Pain Intensity in the Index Joint From Baseline to 24-72 Hours for the First Gout Flare Treated in the Study as Measured by VAS
Description: Patients will score their pain intensity in the joint most affected at baseline (index joint) on a 0-100 mm visual analogue scale (VAS), ranging from no pain (0) to unbearable pain (100). Average of the assessments performed at 24, 48 and 72 hours.
Time Frame: At baseline (pre-dose) and at 24, 48 and 72 hours for the first gout flare treated in the study
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
Units on a scale
  24 hours | -26.1 [-32.5 to -19.6] | -32.5 [-38.8 to -26.1] | -31.1 [-37.6 to -24.6]
  48 hours | -43.4 [-50.8 to -36.0] | -42.9 [-50.0 to -35.9] | -43.6 [-51.0 to -36.3]
  72 hours | -45.2 [-52.7 to -37.7] | -51.6 [-58.9 to -44.3] | -49.1 [-56.5 to -41.6]

2. Secondary Outcome: Change in Patient-assessed Pain Intensity in the Index Joint From Baseline at Time Points From 6 Hours to 8 Days for the First Gout Flare Treated in the Study as Measured by 5-point Likert Scale
Description: Patients will score their pain intensity in the joint most affected at baseline (index joint) on a 5-point Likert scale (0-4 point scale: "none", "mild", "moderate", "severe", "extreme") at time points baseline (pre-dose) and at 6, 12, 18, 24, 36, 48 and 72 hours and Day 5, 6, 7 and 8.
Time Frame: At baseline (pre-dose) and at 6, 12, 18, 24, 36, 48 and 72 hours and Day 5, 6, 7 and 8 for the first gout flare treated in the study
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
Score on a scale
  6 hours | -0.6 (0.7) | -0.8 (0.9) | -0.4 (0.8)
  12 hours | -0.9 (0.6) | -1.1 (1.2) | -0.5 (0.7)
  18 hours | -0.8 (0.8) | -1.2 (1.0) | -0.8 (0.9)
  24 hours | -1.0 (0.8) | -0.9 (1.0) | -1.1 (0.9)
  36 hours | -1.3 (0.8) | -1.3 (1.0) | -1.1 (0.7)
  48 hours | -1.5 (1.0) | -1.4 (1.0) | -1.5 (1.0)
  72 hours | -1.6 (1.1) | -1.6 (1.0) | -1.7 (0.9)
  Day 5 | -1.8 (1.1) | -1.8 (1.1) | -1.8 (1.1)
  Day 6 | -1.9 (1.1) | -2.2 (1.1) | -1.9 (1.0)
  Day 7 | -2.4 (0.8) | -2.2 (1.1) | -1.9 (1.0)
  Day 8 | -1.9 (0.9) | -2.1 (1.1) | -2.1 (1.0)

3. Secondary Outcome: Median Time to Onset of Effect
Description: Onset of effect defined as 20% change from baseline pain intensity in the index joint on a visual analogue scale (VAS)
Time Frame: From baseline (predose) up to Day15 of the first flare treated in the study
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
Hours | 22.3 [13.9 to 24.6] | 11.8 [7.7 to 24.0] | 19.8 [12.1 to 30.0]

4. Secondary Outcome: Median Time to Response
Description: Response defined as 50% change from baseline pain intensity on a visual analogue scale (VAS)
Time Frame: From baseline (predose) up to Day15 of the first flare treated in the study
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
Hours | 47.6 [40.3 to 67.7] | 43.0 [18.6 to 70.4] | 46.9 [24.1 to 67.4]

5. Secondary Outcome: Median Time to Resolution of Pain
Description: Resolution of pain defined as <10 mm on VAS, a continuous 0 to 100 mm visual analogue scale, ranging from no pain (0) to unbearable pain (100), in the index joint
Time Frame: From baseline (predose) up to Day15 of the first flare
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
Hours | 167.5 [120.1 to 264.2] | 131.8 [70.9 to NA] — SAS Proc Lifetest was used. Abridged explanation from the SAS documentation: "Consider the linear transform [..] If the curve that represents the upper confidence limits lies above 0.75, the upper confidence limit for Q1 cannot be estimated[..]." | 119.8 [69.0 to 144.2]

6. Secondary Outcome: Median Time to First Intake of Rescue Medication From First Investigational Drug Administration
Description: Time to first intake of rescue medication for acute gout, measured in hours from first investigational drug administration
Time Frame: From Day 1 to Day 15 for the first flare treated
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 25 | 26 | 22
Hours | NA [126.5 to NA] — Non-calculable | NA [114.4 to NA] — Non-calculable | NA [220.7 to NA] — Non-calculable

7. Secondary Outcome: Physician's Assessment of Global Response to Treatment
Description: 5-point Likert scale (0- to 4-point scale: "none", "mild", "moderate", "severe, "extreme") where higher score mean worse outcome
Time Frame: At 72 hours, Day 8 and Day 15 for the first flare treated in the study
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
Score on a scale
  72 hours | 1.54 [1.23 to 1.85] | 1.25 [0.94 to 1.55] | 1.25 [0.94 to 1.56]
  Day 8 | 1.26 [0.93 to 1.59] | 0.90 [0.59 to 1.20] | 0.81 [0.48 to 1.14]
  Day 15 | 1.04 [0.69 to 1.39] | 0.80 [0.47 to 1.13] | 0.78 [0.46 to 1.13]

8. Secondary Outcome: Physician's Assessment of Clinical Signs in Index Joint: Tenderness
Description: 4-point Likert scale (0=no pain, 1= mild/patient states there is pain when touched, 2= moderate/patient states there is pain and Winces, 3=severe/patient states there is pain, winces and withdraws
Time Frame: at 72 hours, Day 8 and Day 15 for the first flare treated in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
Participants
  72 hours : None | 8 | 18 | 16
  72 hours : Mild | 22 | 28 | 25
  72 hours : Moderate | 17 | 4 | 9
  72 hours : Severe | 4 | 3 | 1
  72 hours : Missing | 4 | 3 | 3
  Day 8 : None | 19 | 28 | 30
  Day 8 : Mild | 25 | 19 | 17
  Day 8 : Moderate | 4 | 2 | 1
  Day 8 : Severe | 1 | 4 | 1
  Day 8 : Missing | 6 | 3 | 5
  Day 15 : None | 37 | 38 | 32
  Day 15 : Mild | 10 | 9 | 12
  Day 15 : Moderate | 1 | 5 | 5
  Day 15 : Severe | 1 | 1 | 0
  Day 15 : Missing | 6 | 3 | 5

9. Secondary Outcome: Physician's Assessment of Clinical Signs in Index Joint: Swelling
Description: 4-point Likert scale (0=no swelling, 1= mild swelling, 2=moderate swelling, 3=severe swelling or bulging beyond joint margins)
Time Frame: at 72 hours, Day 8 and Day 15 for the first flare treated in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
Participants
  Baseline : None | 0 | 0 | 0
  Baseline : Mild | 9 | 14 | 7
  Baseline : Moderate | 23 | 27 | 28
  Baseline : Severe | 23 | 15 | 18
  Baseline : Missing | 0 | 0 | 1
  72 hours : None | 14 | 27 | 17
  72 hours : Mild | 22 | 18 | 26
  72 hours : Moderate | 10 | 7 | 7
  72 hours : Severe | 5 | 1 | 1
  72 hours : Missing | 4 | 3 | 3
  Day 8 : None | 25 | 37 | 38
  Day 8 : Mild | 16 | 13 | 9
  Day 8 : Moderate | 7 | 2 | 2
  Day 8 : Severe | 1 | 1 | 0
  Day 8 : Missing | 6 | 3 | 5
  Day 15 : None | 37 | 44 | 34
  Day 15 : Mild | 9 | 6 | 14
  Day 15 : Moderate | 2 | 3 | 1
  Day 15 : Severe | 1 | 0 | 0
  Day 15 : Missing | 6 | 3 | 5

10. Secondary Outcome: Physician's Assessment of Clinical Signs in Index Joint: Erythema
Description: Physicians assessment of clinical signs with 2 outcomes: Absent=no erythema, present=erythema
Time Frame: at 72 hours, Day 8 and Day 15 for the first flare treated in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
Participants
  Baseline : Absent | 3 | 8 | 8
  Baseline : Present | 51 | 48 | 45
  Baseline : Missing | 1 | 0 | 1
  72 hours : Absent | 29 | 39 | 37
  72 hours : Present | 22 | 14 | 14
  72 hours : Missing | 4 | 3 | 3
  Day 8 : Absent | 43 | 43 | 40
  Day 8 : Present | 6 | 9 | 9
  Day 8 : Missing | 6 | 4 | 5
  Day 15 : Absent | 47 | 47 | 40
  Day 15 : Present | 2 | 5 | 9
  Day 15 : Missing | 6 | 4 | 5

11. Secondary Outcome: Patient´s Assessment of Global Response to Treatment (5-point Likert Scale)
Description: 5-point Likert scale (0- to 4-point scale: 0=excellent, 1=very good, 2=good, 3=fair, 4=poor response to treatment) where lower rate indicates better response to treatment
Time Frame: at 72 hours, Day 8 and Day 15 for the first flare treated in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
Participants
  72 hours : Excellent | 11 | 10 | 18
  72 hours : Very good | 13 | 19 | 9
  72 hours : Good | 7 | 14 | 15
  72 hours : Fair | 7 | 4 | 3
  72 hours : Poor | 4 | 1 | 1
  72 hours : Missing | 13 | 8 | 8
  Day 8 : Excellent | 9 | 16 | 19
  Day 8 : Very good | 16 | 21 | 13
  Day 8 : Good | 8 | 6 | 7
  Day 8 : Fair | 5 | 6 | 2
  Day 8 : Poor | 5 | 0 | 1
  Day 8 : Missing | 12 | 7 | 12
  Day 15 : Excellent | 14 | 19 | 21
  Day 15 : Very good | 9 | 13 | 11
  Day 15 : Good | 10 | 8 | 10
  Day 15 : Fair | 6 | 5 | 3
  Day 15 : Poor | 3 | 0 | 1
  Day 15 : Missing | 13 | 11 | 8

12. Secondary Outcome: Change From Baseline in the Inflammatory Biomarker C Reactive Protein
Description: This endpoint represents the change from baseline, mg/dL, of the inflammatory biomarker C reactive protein
Time Frame: baseline (predose) and at 72 hours, Day 8 and Day 15 for the first flare treated in the study
Population: Some patients did not undertake all assessments.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
mg/dL
  72 hours: number analyzed (Participants) | 45 | 45 | 45
  72 hours | -0.362 (3.435) | -1.435 (2.057) | -1.362 (1.682)
  Day 8: number analyzed (Participants) | 34 | 40 | 43
  Day 8 | -0.321 (2.153) | -1.334 (2.702) | 1.406 (1.961)
  Day 15: number analyzed (Participants) | 39 | 42 | 38
  Day 15 | -1.102 (1.690) | -0.724 (2.525) | -0.607 (2.646)

13. Secondary Outcome: Change From Baseline in the Inflammatory Biomarker Serum Amyloid A
Description: This endpoint represents the change from baseline, mg/L, of the inflammatory biomarker Serum amyloid A
Time Frame: baseline (predose) and at 72 hours, Day 8 and Day 15 for the first flare treated in the study
Population: Some patients did not undertake all assessments.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
mg/L
  72 hours: number analyzed (Participants) | 43 | 45 | 46
  72 hours | 8.950 (246.317) | -45.160 (126.986) | -34.510 (58.518)
  Day 8: number analyzed (Participants) | 36 | 41 | 42
  Day 8 | -6.363 (117.794) | -46.561 (144.630) | -35.887 (64.144)
  Day 15: number analyzed (Participants) | 40 | 39 | 39
  Day 15 | -50.524 (105.170) | -25.328 (144.039) | 14.370 (146.627)

14. Secondary Outcome: The Percent of Patients With at Least One Adverse Event
Description: All adverse events to be recorded Day 1 - Day 28 for each flare. Serious adverse events (SAE) will be collected from informed consent until week 12 for each flare. Any SAE with suspected causal relationship should be reported irrespective of the time of occurrence.
Time Frame: Through study completion, at 12 weeks after last flare treated during the extension period
Measure: Number; unit: Percent
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 54 | 55 | 52
Percent | 40.7 | 38.2 | 55.8

15. Secondary Outcome: The Percent of Patients With at Least One Serious Adverse Event, Including Death
Description: Serious Adverse Events (SAE) will be collected from informed consent until week 12 for each flare. Any SAE with suspected causal relationship should be reported irrespective of the time of occurrence.
Time Frame: Through study completion, at 12 weeks after last flare treated during the extension period
Measure: Number; unit: Percent
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 54 | 55 | 52
Percent | 0 | 7.3 | 0

16. Secondary Outcome: Serum Concentration of Endogenous Interleukin-1 Receptor Antagonist /Anakinra
Description: This endpoint represents the level of of endogenous interleukin-1 receptor antagonist /anakinra
Time Frame: Baseline (predose) and at 72 hours, Day 8, Day 15, Day 28 and Week 12 for the first flare and subsequent flares treated during the extension period
Population: Some patients did not undertake all assessments.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 54 | 55 | 52
ng/mL
  First flare : Baseline: number analyzed (Participants) | 51 | 53 | 51
  First flare : Baseline | 2.032 (2.493) | 4.883 (24.378) | 1.950 (2.755)
  First flare : 72 hours: number analyzed (Participants) | 49 | 54 | 51
  First flare : 72 hours | 1.974 (1.793) | 267.744 (246.086) | 628.053 (540.488)
  First flare : Day 8: number analyzed (Participants) | 49 | 54 | 49
  First flare : Day 8 | 1.692 (1.343) | 6.750 (10.439) | 34.777 (87.812)
  First flare : Day 15: number analyzed (Participants) | 47 | 51 | 47
  First flare : Day 15 | 1.533 (0.226) | 1.588 (0.443) | 1.574 (0.356)
  First flare : Day 28: number analyzed (Participants) | 40 | 44 | 39
  First flare : Day 28 | 1.635 (0.615) | 1.659 (1.057) | 1.779 (0.895)
  First flare : Week 12: number analyzed (Participants) | 32 | 30 | 30
  First flare : Week 12 | 1.500 (0.000) | 1.625 (0.478) | 1.719 (0.681)
  Second flare : Baseline: number analyzed (Participants) | 17 | 23 | 21
  Second flare : Baseline | 1.748 (1.024) | 1.718 (0.732) | 1.500 (0.00)
  Second flare : 72 hours: number analyzed (Participants) | 17 | 21 | 21
  Second flare : 72 hours | 1.628 (0.526) | 254.930 (249.962) | 719.667 (840.530)
  Second flare : Day 8: number analyzed (Participants) | 17 | 22 | 21
  Second flare : Day 8 | 3.141 (6.270) | 7.048 (20.338) | 48.785 (114.114)
  Second flare : Day 15: number analyzed (Participants) | 14 | 23 | 20
  Second flare : Day 15 | 1.845 (1291) | 1.595 (0.457) | 1.500 (0.00)
  Second flare : Day 28: number analyzed (Participants) | 13 | 21 | 14
  Second flare : Day 28 | 1.975 (1.714) | 1.692 (0.882) | 1.500 (0.00)
  Second flare : Week 12: number analyzed (Participants) | 10 | 16 | 11
  Second flare : Week 12 | 2.920 (4.490) | 1.681 (0.725) | 1.692 (0.636)
  Third flare : Baseline: number analyzed (Participants) | 15 | 13 | 13
  Third flare : Baseline | 2.05 (1.24) | 1.50 (0.00) | 1.50 (0.00)
  Third flare : 72 hours: number analyzed (Participants) | 5 | 13 | 12
  Third flare : 72 hours | 1.85 (0.78) | 196.67 (192.56) | 431.63 (298.51)
  Third flare : Day 8: number analyzed (Participants) | 5 | 12 | 11
  Third flare : Day 8 | 1.50 (0.00) | 5.56 (12.97) | 10.70 (15.42)
  Third flare : Day 15: number analyzed (Participants) | 5 | 12 | 11
  Third flare : Day 15 | 1.50 (0.00) | 1.63 (0.44) | 1.50 (0.00)
  Third flare : Day 28: number analyzed (Participants) | 5 | 10 | 6
  Third flare : Day 28 | 1.85 (0.78) | 1.50 (0.00) | 2.47 (2.38)
  Third flare : Week 12: number analyzed (Participants) | 2 | 9 | 3
  Third flare : Week 12 | 2.85 (1.91) | 1.50 (0.00) | 1.50 (0.00)
  Fourth flare : Baseline: number analyzed (Participants) | 3 | 7 | 10
  Fourth flare : Baseline | 1.50 (0.00) | 1.50 (0.00) | 1.50 (0.00)
  Fourth flare : 72 hours: number analyzed (Participants) | 3 | 6 | 9
  Fourth flare : 72 hours | 1.50 (0.00) | 184.40 (198.19) | 916.62 (1549.55)
  Fourth flare : Day 8: number analyzed (Participants) | 3 | 7 | 10
  Fourth flare : Day 8 | 1.50 (0.00) | 1.89 (1.02) | 20.62 (34.10)
  Fourth flare : Day 15: number analyzed (Participants) | 3 | 7 | 9
  Fourth flare : Day 15 | 1.50 (0.00) | 1.50 (0.00) | 1.50 (0.00)
  Fourth flare : Day 28: number analyzed (Participants) | 2 | 5 | 7
  Fourth flare : Day 28 | 1.50 (0.00) | 1.50 (0.00) | 1.50 (0.00)
  Fourth flare : Week 12: number analyzed (Participants) | 1 | 5 | 3
  Fourth flare : Week 12 | 1.50 (0.00) | 2.66 (2.60) | 1.50 (0.00)
  Fifth flare : Baseline: number analyzed (Participants) | 3 | 3 | 6
  Fifth flare : Baseline | 1.50 (0.00) | 1.50 (0.00) | 1.50 (0.00)
  Fifthe flare : 72 hours: number analyzed (Participants) | 3 | 3 | 6
  Fifthe flare : 72 hours | 1.50 (0.00) | 129.20 (200.26) | 292.35 (308.56)
  Fifthe flare : Day 8: number analyzed (Participants) | 3 | 3 | 6
  Fifthe flare : Day 8 | 1.50 (0.00) | 1.50 (0.00) | 6.39 (9.49)
  Fifthe flare : Day 15: number analyzed (Participants) | 3 | 3 | 6
  Fifthe flare : Day 15 | 1.50 (0.00) | 1.50 (0.00) | 1.50 (0.00)
  Fifthe flare : Day 28: number analyzed (Participants) | 3 | 2 | 6
  Fifthe flare : Day 28 | 1.50 (0.00) | 3.31 (2.55) | 1.50 (0.00)
  Fifth flare : Week 12: number analyzed (Participants) | 2 | 0 | 5
  Fifth flare : Week 12 | 1.50 (0.00) |  | 1.50 (0.00)

17. Secondary Outcome: Proportion of Patients With Anti-drug Antibodies (ADA) Against Anakinra
Description: Confirmed ADA positive samples will be analysed for the presence of neutralizing antibodies
Time Frame: Baseline (predose) and at 72 hours, Day 8, Day 15, Day 28 and Week 12 for the first flare and subsequent flares treated treated during the extension period
Population: Some patients did not undertake all assessments.
Measure: Number; unit: participants
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 54 | 55 | 52
participants
  First flare : Baseline | 2 | 5 | 2
  First flare : Day 8 | 1 | 4 | 3
  First flare : Day 15 | 0 | 5 | 4
  First flare : Day 28 | 0 | 4 | 2
  First flare : Week 12 | 0 | 4 | 0
  Second flare : Baseline: number analyzed (Participants) | 17 | 23 | 21
  Second flare : Baseline | 0 | 0 | 2
  Second flare : Day 8: number analyzed (Participants) | 17 | 23 | 21
  Second flare : Day 8 | 0 | 1 | 2
  Second flare : Day 15: number analyzed (Participants) | 17 | 23 | 21
  Second flare : Day 15 | 0 | 1 | 0
  Second flare : Day 28: number analyzed (Participants) | 17 | 23 | 21
  Second flare : Day 28 | 0 | 1 | 1
  Second flare : Week 12: number analyzed (Participants) | 17 | 23 | 21
  Second flare : Week 12 | 0 | 0 | 1
  Third flare : Baseline: number analyzed (Participants) | 5 | 13 | 13
  Third flare : Baseline | 0 | 0 | 2
  Third flare : Day 8: number analyzed (Participants) | 5 | 13 | 13
  Third flare : Day 8 | 0 | 1 | 4
  Third flare : Day 15: number analyzed (Participants) | 5 | 13 | 13
  Third flare : Day 15 | 0 | 1 | 4
  Third flare : Day 28: number analyzed (Participants) | 5 | 13 | 13
  Third flare : Day 28 | 0 | 1 | 0
  Third flare : Week 12: number analyzed (Participants) | 5 | 13 | 13
  Third flare : Week 12 | 0 | 0 | 0
  Fourth flare : Baseline: number analyzed (Participants) | 3 | 7 | 10
  Fourth flare : Baseline | 0 | 0 | 2
  Fourth flare : Day 8: number analyzed (Participants) | 3 | 7 | 10
  Fourth flare : Day 8 | 0 | 1 | 3
  Fourth flare : Day 15: number analyzed (Participants) | 3 | 7 | 10
  Fourth flare : Day 15 | 0 | 1 | 4
  Fourth flare : Day 28: number analyzed (Participants) | 3 | 7 | 10
  Fourth flare : Day 28 | 0 | 1 | 1
  Fourth flare : Week 12: number analyzed (Participants) | 3 | 7 | 10
  Fourth flare : Week 12 | 0 | 1 | 0
  Fifth flare : Baseline: number analyzed (Participants) | 3 | 3 | 6
  Fifth flare : Baseline | 0 | 0 | 1
  Fifth flare : Day 8: number analyzed (Participants) | 3 | 3 | 6
  Fifth flare : Day 8 | 0 | 1 | 2
  Fifth flare : Day 15: number analyzed (Participants) | 3 | 3 | 6
  Fifth flare : Day 15 | 0 | 2 | 2
  Fifth flare : Day 28: number analyzed (Participants) | 3 | 3 | 6
  Fifth flare : Day 28 | 0 | 1 | 2
  Fifth flare : Week 12: number analyzed (Participants) | 3 | 3 | 6
  Fifth flare : Week 12 | 0 | 0 | 0

18. Secondary Outcome: Proportion of Patients With Neutralizing Antibodies
Description: Confirmed ADA positive samples will be analysed for the presence of neutralizing antibodies
Time Frame: as for outcome 16
Population: Some patients did not undertake all assessments.
Measure: Number; unit: participants
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 54 | 55 | 52
participants
  First flare : Baseline | 0 | 0 | 0
  First flare : Day 8 | 0 | 0 | 0
  First flare : Day 15 | 0 | 0 | 0
  First flare : Day 28 | 0 | 0 | 0
  First flare : Week 12 | 0 | 0 | 0
  Second flare : Study baseline: number analyzed (Participants) | 17 | 23 | 21
  Second flare : Study baseline | 0 | 0 | 0
  Second flare : Flare baseline: number analyzed (Participants) | 17 | 23 | 21
  Second flare : Flare baseline | 0 | 0 | 0
  Second flare : Day 8: number analyzed (Participants) | 17 | 23 | 21
  Second flare : Day 8 | 0 | 0 | 0
  Second flare : Day 15: number analyzed (Participants) | 17 | 23 | 21
  Second flare : Day 15 | 0 | 0 | 0
  Second flare : Day 28: number analyzed (Participants) | 17 | 23 | 21
  Second flare : Day 28 | 0 | 0 | 0
  Second flare : Week 12: number analyzed (Participants) | 17 | 23 | 21
  Second flare : Week 12 | 0 | 0 | 0
  Third flare : Study baseline: number analyzed (Participants) | 5 | 13 | 13
  Third flare : Study baseline | 0 | 0 | 0
  Third flare : Flare baseline: number analyzed (Participants) | 5 | 13 | 13
  Third flare : Flare baseline | 0 | 0 | 0
  Third flare : Day 8: number analyzed (Participants) | 5 | 13 | 13
  Third flare : Day 8 | 0 | 0 | 0
  Third flare : Day 15: number analyzed (Participants) | 5 | 13 | 13
  Third flare : Day 15 | 0 | 0 | 0
  Third flare : Day 28: number analyzed (Participants) | 5 | 13 | 13
  Third flare : Day 28 | 0 | 0 | 0
  Third flare : Week 12: number analyzed (Participants) | 5 | 13 | 13
  Third flare : Week 12 | 0 | 0 | 0
  Fourth flare : Study baseline: number analyzed (Participants) | 3 | 7 | 10
  Fourth flare : Study baseline | 0 | 0 | 0
  Fourth flare : Flare baseline: number analyzed (Participants) | 3 | 7 | 10
  Fourth flare : Flare baseline | 0 | 0 | 0
  Fourth flare : Day 8: number analyzed (Participants) | 3 | 7 | 10
  Fourth flare : Day 8 | 0 | 1 | 0
  Fourth flare : Day 15: number analyzed (Participants) | 3 | 7 | 10
  Fourth flare : Day 15 | 0 | 0 | 1
  Fourth flare : Day 28: number analyzed (Participants) | 3 | 7 | 10
  Fourth flare : Day 28 | 0 | 0 | 0
  Fourth flare : Week 12: number analyzed (Participants) | 3 | 7 | 10
  Fourth flare : Week 12 | 0 | 0 | 0
  Fifth flare : Study baseline: number analyzed (Participants) | 3 | 3 | 6
  Fifth flare : Study baseline | 0 | 0 | 0
  Fifth flare : Flare baseline: number analyzed (Participants) | 3 | 3 | 6
  Fifth flare : Flare baseline | 0 | 0 | 0
  Fifth flare : Day 8: number analyzed (Participants) | 3 | 3 | 6
  Fifth flare : Day 8 | 0 | 0 | 0
  Fifth flare : Day 15: number analyzed (Participants) | 3 | 3 | 6
  Fifth flare : Day 15 | 0 | 0 | 0
  Fifth flare : Day 28: number analyzed (Participants) | 3 | 3 | 6
  Fifth flare : Day 28 | 0 | 0 | 0
  Fifth flare : Week 12: number analyzed (Participants) | 3 | 3 | 6
  Fifth flare : Week 12 | 0 | 0 | 0

19. Secondary Outcome: Change From Baseline in Short Form (36) Health Survey, Acute Version 2 (SF-36®) Physical Functioning Domain Score
Description: SF-36® measures the impact of disease on overall quality of life. It consists of 8 individual domains. Score range from 0 to 100, where 0 represents the worst possible health and 100 is perfect health.
Time Frame: at baseline, Day 8 and Day 15 for the first flare treated in the study
Population: Some patients did not undertake all assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
units on a scale
  Day 8: number analyzed (Participants) | 42 | 47 | 40
  Day 8 | 8.0 (9.8) | 10.5 (10.0) | 10.4 (8.3)
  Day 15: number analyzed (Participants) | 39 | 44 | 44
  Day 15 | 11.8 (8.2) | 12.2 (11.9) | 9.4 (8.7)

20. Secondary Outcome: Change From Baseline in Health Related Quality of Life EuroQol 5 Dimensions 5 Levels (EQ-5D-5L)
Description: Exploratory objective. The EQ-5D-5L, a self-report questionnaire, is a descriptive system of Health related quality of life (HRQL) states consisting of 5 dimensions (Mobility, Self-care, Usual activities, Pain/Discomfort, Anxiety/Depression), each of which can have 5 responses. The responses record 5 levels of severity (no problems/slight problems/moderate problems/severe problems/extreme problems) within a particular EQ-5D dimension.
Time Frame: at baseline, Day 8 and Day 15 for the first flare treated in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
Participants
  Mobility scores : Day 8: Improvement 4 step | 2 | 1 | 0
  Mobility scores : Day 8: Improvement 3 step | 5 | 6 | 5
  Mobility scores : Day 8: Improvement 2 step | 12 | 9 | 11
  Mobility scores : Day 8: Improvement 1 step | 5 | 18 | 12
  Mobility scores : Day 8: No change | 14 | 7 | 9
  Mobility scores : Day 8: Deterioration 1 steps | 3 | 3 | 2
  Mobility scores : Day 8: Deterioration 2 steps | 0 | 3 | 0
  Mobility scores : Day 8: Deterioration 3 steps | 0 | 0 | 0
  Mobility scores : Day 8: Detorioration 4 steps | 0 | 0 | 0
  Mobility scores : Day 8: Missing | 14 | 9 | 15
  Mobility scores : Day 15: Improvement 4 step | 2 | 1 | 0
  Mobility scores : Day 15: Improvement 3 step | 7 | 7 | 2
  Mobility scores : Day 15: Improvement 2 step | 11 | 10 | 15
  Mobility scores : Day 15: Improvement 1 step | 8 | 16 | 10
  Mobility scores : Day 15: No change | 9 | 5 | 14
  Mobility scores : Day 15: Deterioration 1 steps | 1 | 4 | 2
  Mobility scores : Day 15: Deterioration 2 steps | 0 | 1 | 0
  Mobility scores : Day 15: Deterioration 3 steps | 0 | 0 | 0
  Mobility scores : Day 15: Detorioration 4 steps | 0 | 0 | 0
  Mobility scores : Day 15: Missing | 17 | 12 | 11
  Self-care scores : Day 8: Improvement 4 step | 2 | 1 | 0
  Self-care scores : Day 8: Improvement 3 step | 3 | 3 | 3
  Self-care scores : Day 8: Improvement 2 step | 4 | 3 | 7
  Self-care scores : Day 8: Improvement 1 step | 7 | 11 | 6
  Self-care scores : Day 8: No change | 23 | 27 | 22
  Self-care scores : Day 8: Deterioration 1 steps | 1 | 1 | 1
  Self-care scores : Day 8: Deterioration 2 steps | 1 | 1 | 0
  Self-care scores : Day 8: Deterioration 3 steps | 0 | 0 | 0
  Self-care scores : Day 8: Detorioration 4 steps | 0 | 0 | 0
  Self-care scores : Day 8: Missing | 14 | 9 | 15
  Selfcare scores : Day 15: Improvement 4 step | 2 | 1 | 0
  Selfcare scores : Day 15: Improvement 3 step | 2 | 3 | 1
  Selfcare scores : Day 15: Improvement 2 step | 5 | 5 | 7
  Selfcare scores : Day 15: Improvement 1 step | 8 | 10 | 10
  Selfcare scores : Day 15: No change | 20 | 21 | 25
  Selfcare scores : Day 15: Deterioration 1 steps | 1 | 3 | 0
  Selfcare scores : Day 15: Deterioration 2 steps | 0 | 1 | 0
  Selfcare scores : Day 15: Deterioration 3 steps | 0 | 0 | 0
  Selfcare scores : Day 15: Detorioration 4 steps | 0 | 0 | 0
  Selfcare scores : Day 15: Missing | 17 | 12 | 11
  Usual activities scores : Day 8: Improvement 4 step | 3 | 0 | 0
  Usual activities scores : Day 8: Improvement 3 step | 3 | 6 | 2
  Usual activities scores : Day 8: Improvement 2 step | 15 | 11 | 13
  Usual activities scores : Day 8: Improvement 1 step | 10 | 14 | 9
  Usual activities scores : Day 8: No change | 6 | 12 | 14
  Usual activities scores : Day 8: Deterioration 1 steps | 4 | 2 | 1
  Usual activities scores : Day 8: Deterioration 2 steps | 0 | 2 | 0
  Usual activities scores : Day 8: Deterioration 3 steps | 0 | 0 | 0
  Usual activities scores : Day 8: Detorioration 4 steps | 0 | 0 | 0
  Usual activities scores : Day 8: Missing | 14 | 9 | 15
  Usual activities scores : Day 15: Improvement 4 step | 2 | 1 | 0
  Usual activities scores : Day 15: Improvement 3 step | 8 | 7 | 0
  Usual activities scores : Day 15: Improvement 2 step | 10 | 11 | 13
  Usual activities scores : Day 15: Improvement 1 step | 10 | 12 | 13
  Usual activities scores : Day 15: No change | 6 | 9 | 14
  Usual activities scores : Day 15: Deterioration 1 steps | 2 | 3 | 2
  Usual activities scores : Day 15: Deterioration 2 steps | 0 | 1 | 1
  Usual activities scores : Day 15: Deterioration 3 steps | 0 | 0 | 0
  Usual activities scores : Day 15: Detorioration 4 steps | 0 | 0 | 0
  Usual activities scores : Day 15: Missing | 17 | 12 | 11
  Pain/discomfort scores : Day 8: Improvement 4 step | 3 | 3 | 0
  Pain/discomfort scores : Day 8: Improvement 3 step | 5 | 11 | 11
  Pain/discomfort scores : Day 8: Improvement 2 step | 16 | 12 | 15
  Pain/discomfort scores : Day 8: Improvement 1 step | 12 | 15 | 9
  Pain/discomfort scores : Day 8: No change | 4 | 4 | 4
  Pain/discomfort scores : Day 8: Deterioration 1 steps | 0 | 1 | 0
  Pain/discomfort scores : Day 8: Deterioration 2 steps | 1 | 1 | 0
  Pain/discomfort scores : Day 8: Deterioration 3 steps | 0 | 0 | 0
  Pain/discomfort scores : Day 8: Detorioration 4 steps | 0 | 0 | 0
  Pain/discomfort scores : Day 8: Missing | 14 | 9 | 15
  Pain/discomfort scores : Day 15: Improvement 4 step | 3 | 3 | 1
  Pain/discomfort scores : Day 15: Improvement 3 step | 9 | 11 | 10
  Pain/discomfort scores : Day 15: Improvement 2 step | 17 | 13 | 14
  Pain/discomfort scores : Day 15: Improvement 1 step | 5 | 11 | 10
  Pain/discomfort scores : Day 15: No change | 3 | 2 | 8
  Pain/discomfort scores : Day 15: Deterioration 1 steps | 1 | 3 | 0
  Pain/discomfort scores : Day 15: Deterioration 2 steps | 0 | 1 | 0
  Pain/discomfort scores : Day 15: Deterioration 3 steps | 0 | 0 | 0
  Pain/discomfort scores : Day 15: Detorioration 4 steps | 0 | 0 | 0
  Pain/discomfort scores : Day 15: Missing | 17 | 12 | 11
  Anxiety/depression scores : Day 8: Improvement 4 step | 1 | 0 | 0
  Anxiety/depression scores : Day 8: Improvement 3 step | 2 | 2 | 0
  Anxiety/depression scores : Day 8: Improvement 2 step | 3 | 0 | 3
  Anxiety/depression scores : Day 8: Improvement 1 step | 5 | 9 | 9
  Anxiety/depression scores : Day 8: No change | 26 | 33 | 25
  Anxiety/depression scores : Day 8: Deterioration 1 steps | 4 | 3 | 2
  Anxiety/depression scores : Day 8: Deterioration 2 steps | 0 | 0 | 0
  Anxiety/depression scores : Day 8: Deterioration 3 steps | 0 | 0 | 0
  Anxiety/depression scores : Day 8: Detorioration 4 steps | 0 | 0 | 0
  Anxiety/depression scores : Day 8: Missing | 14 | 9 | 15
  Anxiety/depression scores : Day 15: Improvement 4 step | 1 | 0 | 0
  Anxiety/depression scores : Day 15: Improvement 3 step | 1 | 2 | 0
  Anxiety/depression scores : Day 15: Improvement 2 step | 4 | 1 | 3
  Anxiety/depression scores : Day 15: Improvement 1 step | 7 | 6 | 10
  Anxiety/depression scores : Day 15: No change | 23 | 33 | 26
  Anxiety/depression scores : Day 15: Deterioration 1 steps | 0 | 2 | 4
  Anxiety/depression scores : Day 15: Deterioration 2 steps | 2 | 0 | 0
  Anxiety/depression scores : Day 15: Deterioration 3 steps | 0 | 0 | 0
  Anxiety/depression scores : Day 15: Detorioration 4 steps | 0 | 0 | 0
  Anxiety/depression scores : Day 15: Missing | 17 | 12 | 11

21. Secondary Outcome: Percent Impairment While Working During Last Week Due to Gout During the First Flare and Subsequent Flares
Description: The WPAI yeilds four types of scores of which Work productivity loss is one.
  SHP is derived from WPAI as follows:
  The WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity as follows:
  Questions:
  Q1 = currently employed Q2 = hours missed due to specified problem Q3 = hours missed other reasons Q4 = hours actually worked Q5 = degree problem affected productivity while working Q6 = degree problem affected regular activities
  Scores:
  Multiply scores by 100 to express in percentages. Percent impairment while working due to problem: Q5/10 The answer on Q5 is given on a scale from 0 (PROBLEM had no effect on work) to 10 (PROBLEM completely prevented me from working).
  Thus the analysis values from which mean and SD have been calculated and reported are the outcomes from Q5 (ranging from 0 to 10) multiplied with 100 and divided by 10.
Time Frame: Recorded up to Day 15 for the first flare and subsequent flares treated during the extension period
Population: Some patients did not undertake all assessments.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
percent
  First flare : Day 8: number analyzed (Participants) | 18 | 23 | 19
  First flare : Day 8 | 36.1 (34.3) | 32.6 (29.1) | 20.5 (25.0)
  First flare : Day 15: number analyzed (Participants) | 21 | 23 | 25
  First flare : Day 15 | 23.3 (24.8) | 12.6 (20.7) | 21.6 (22.3)
  Second flare : Day 8: number analyzed (Participants) | 7 | 10 | 10
  Second flare : Day 8 | 42.9 (27.5) | 24.0 (26.3) | 24.0 (27.2)
  Second flare : Day 15: number analyzed (Participants) | 5 | 10 | 8
  Second flare : Day 15 | 16.0 (25.1) | 20.0 (17.6) | 13.8 (16.9)
  Third flare : Day 8: number analyzed (Participants) | 1 | 2 | 3
  Third flare : Day 8 | 10.0 | 5.0 (7.1) | 10.0 (10.0)
  Third flare : Day 15: number analyzed (Participants) | 1 | 4 | 3
  Third flare : Day 15 | 10.0 | 20.0 (24.5) | 23.3 (32.1)
  Fourth flare : Day 8: number analyzed (Participants) | 1 | 0 | 3
  Fourth flare : Day 8 | 30.0 |  | 20.0 (34.6)
  Fourth flare : Day 15: number analyzed (Participants) | 0 | 0 | 2
  Fourth flare : Day 15 |  |  | 5.0 (7.1)
  Fifth flare : Day 8: number analyzed (Participants) | 1 | 0 | 3
  Fifth flare : Day 8 | 60.0 |  | 26.7 (25.2)
  Fifth flare : Day 15: number analyzed (Participants) | 1 | 1 | 3
  Fifth flare : Day 15 | 20.0 | 40.0 | 13.3 (11.5)

22. Secondary Outcome: Health Care Resource Utilization Due to a Gouty Arthritis Flare
Description: Exploratory objective: number of days with hospitalization and un-scheduled outpatient visits
Time Frame: Recorded up to Day 15 for the first flare and subsequent flares treated during the extension period
Population: Some patients did not undertake all assessments.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
Number analyzed (Participants) | 55 | 56 | 54
days
  Hospitalization : First flare : Day 1-7 | 0 (0) | 0 (0) | 0 (0)
  Hospitalization : First flare : Day 8-15 | 0 (0) | 0 (0) | 0 (0)
  Hospitalization : First flare : Day 1-15 | 0 (0) | 0 (0) | 0 (0)
  Hospitalization : Second flare : Day 1-7: number analyzed (Participants) | 17 | 23 | 21
  Hospitalization : Second flare : Day 1-7 | 0 (0) | 0 (0) | 0 (0)
  Hospitalization : Second flare : Day 8-15: number analyzed (Participants) | 17 | 23 | 21
  Hospitalization : Second flare : Day 8-15 | 0 (0) | 0 (0) | 0 (0)
  Hospitalization : Second flare : Day 1-15: number analyzed (Participants) | 17 | 23 | 21
  Hospitalization : Second flare : Day 1-15 | 0 (0) | 0 (0) | 0 (0)
  Hospitalization : Third flare : Day 1-7: number analyzed (Participants) | 5 | 13 | 13
  Hospitalization : Third flare : Day 1-7 | 0 (0) | 0 (0) | 0 (0)
  Hospitalization : Third flare : Day 8-15: number analyzed (Participants) | 5 | 13 | 13
  Hospitalization : Third flare : Day 8-15 | 0 (0) | 0 (0) | 0 (0)
  Hospitalization : Third flare : Day 1-15: number analyzed (Participants) | 5 | 13 | 13
  Hospitalization : Third flare : Day 1-15 | 0 (0) | 0 (0) | 0 (0)
  Hospitalization : Fourth flare : Day 1-7: number analyzed (Participants) | 3 | 7 | 10
  Hospitalization : Fourth flare : Day 1-7 | 0 (0) | 0 (0) | 0 (0)
  Hospitalization : Fourth flare : Day 8-15: number analyzed (Participants) | 3 | 7 | 10
  Hospitalization : Fourth flare : Day 8-15 | 0 (0) | 0 (0) | 0 (0)
  Hospitalization : Fourth flare : Day 1-15: number analyzed (Participants) | 3 | 7 | 10
  Hospitalization : Fourth flare : Day 1-15 | 0 (0) | 0 (0) | 0 (0)
  Hospitalization : Fifth flare : Day 1-7: number analyzed (Participants) | 3 | 3 | 6
  Hospitalization : Fifth flare : Day 1-7 | 0 (0) | 0 (0) | 0 (0)
  Hospitalization : Fifth flare : Day 8-15: number analyzed (Participants) | 3 | 3 | 6
  Hospitalization : Fifth flare : Day 8-15 | 0 (0) | 0 (0) | 0 (0)
  Hospitalization : Fifth flare : Day 1-15: number analyzed (Participants) | 3 | 3 | 6
  Hospitalization : Fifth flare : Day 1-15 | 0 (0) | 0 (0) | 0 (0)
  Unscheduled outpatient visits:First flare: Day 1-7 | 0.1 (0.5) | 0 (0) | 0.1 (0.6)
  Unscheduled outpatient visits:First flare:Day 8-15 | 0.3 (1.4) | 0.1 (0.6) | 0 (0)
  Unscheduled outpatient visits:First flare:Day 1-15 | 0.4 (1.4) | 0.1 (0.6) | 0.1 (0.6)
  Unscheduled outpatient visits:Second flare:Day 1-7: number analyzed (Participants) | 17 | 23 | 21
  Unscheduled outpatient visits:Second flare:Day 1-7 | 0.2 (0.8) | 0 (0) | 0 (0)
  Unscheduled outpatient visit:Second flare:Day 8-15: number analyzed (Participants) | 17 | 23 | 21
  Unscheduled outpatient visit:Second flare:Day 8-15 | 0.2 (0.6) | 0 (0) | 0 (0)
  Unscheduled outpatient visit:Second flare:Day 1-15: number analyzed (Participants) | 17 | 23 | 21
  Unscheduled outpatient visit:Second flare:Day 1-15 | 0.5 (1.5) | 0 (0) | 0 (0)
  Unscheduled outpatient visits:Third flare:Day 1-7: number analyzed (Participants) | 5 | 13 | 13
  Unscheduled outpatient visits:Third flare:Day 1-7 | 0.4 (0.9) | 0 (0) | 0 (0)
  Unscheduled outpatient visits:Third flare:Day 8-15: number analyzed (Participants) | 5 | 13 | 13
  Unscheduled outpatient visits:Third flare:Day 8-15 | 0.4 (0.9) | 0 (0) | 0 (0)
  Unscheduled outpatient visits:Third flare:Day 1-15: number analyzed (Participants) | 5 | 13 | 13
  Unscheduled outpatient visits:Third flare:Day 1-15 | 0.8 (1.8) | 0 (0) | 0 (0)
  Unscheduled outpatient visitstFourth flare:Day 1-7: number analyzed (Participants) | 3 | 7 | 10
  Unscheduled outpatient visitstFourth flare:Day 1-7 | 0 (0) | 0 (0) | 0 (0)
  Unscheduled outpatient visitsFourth flare:Day 8-15: number analyzed (Participants) | 3 | 7 | 10
  Unscheduled outpatient visitsFourth flare:Day 8-15 | 0 (0) | 0 (0) | 0 (0)
  Unscheduled outpatient visitsFourth flare:Day 1-15: number analyzed (Participants) | 3 | 7 | 10
  Unscheduled outpatient visitsFourth flare:Day 1-15 | 0 (0) | 0 (0) | 0 (0)
  Unscheduled outpatient visit:Fifth flare : Day 1-7: number analyzed (Participants) | 3 | 3 | 6
  Unscheduled outpatient visit:Fifth flare : Day 1-7 | 0 (0) | 0 (0) | 0 (0)
  Unscheduled outpatient visitFifth flare : Day 8-15: number analyzed (Participants) | 3 | 3 | 6
  Unscheduled outpatient visitFifth flare : Day 8-15 | 0 (0) | 0 (0) | 0 (0)
  Unscheduled outpatient visit Fifth flare:Day 1-15: number analyzed (Participants) | 3 | 3 | 6
  Unscheduled outpatient visit Fifth flare:Day 1-15 | 0 (0) | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: The period for recording all adverse events, including SAEs begins upon receiving the first dose of Investigational medicinal product (IMP) and ends with a follow-up telephone call 5 weeks after the first dose of IMP. SAEs will also be collected from signing of the Informed consent form (ICF) until the Week 12 visit
Arm/Group | Triamcinolone 40 mg | Anakinra 100 mg | Anakinra 200 mg
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/55 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/54 | 4/55 | 1/52
Other Adverse Events (participants affected / at risk) | 22/54 | 19/55 | 29/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Triamcinolone 40 mg (N=54) | Anakinra 100 mg (N=55) | Anakinra 200 mg (N=52)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Sickel cell anaemia (Congenital, familial and genetic disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triamcinolone 40 mg (N=54) | Anakinra 100 mg (N=55) | Anakinra 200 mg (N=52)
Influenza (Infections and infestations) | 0 | 3 (3) | 5 (9)
Nasopharyngitis (Infections and infestations) | 0 | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 | 1 (1) | 1 (1)
Escherichia infection (Infections and infestations) | 0 | 0 | 1 (1)
Haemophilus infection (Infections and infestations) | 0 | 0 | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 (1)
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 (1)
Tooth infection (Infections and infestations) | 0 | 0 | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 (1) | 3 (5)
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1 (1) | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 3 (3) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 (0) | 1 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 (1) | 0
Stress (Psychiatric disorders) | 0 | 0 | 1 (2)
Anger (Psychiatric disorders) | 0 | 1 (1) | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 (1)
Mood swings (Psychiatric disorders) | 0 | 1 (1) | 0
Headache (Nervous system disorders) | 2 (2) | 0 | 2 (2)
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 (1)
Nystagmus (Nervous system disorders) | 0 | 0 | 1 (1)
Seizure (Nervous system disorders) | 0 | 0 | 1 (1)
Somnolence (Nervous system disorders) | 0 | 1 (1) | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1) | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 (1) | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 | 0
Flushing (Vascular disorders) | 1 (1) | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 | 1 (1) | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 (1) | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1 (1) | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 (1) | 0
Constipation (Gastrointestinal disorders) | 1 (1) | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 0 | 0 | 2 (2)
Renal failure (Renal and urinary disorders) | 0 | 1 (3) | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 | 0
Type IIa hyperlipidaemia (Congenital, familial and genetic disorders) | 0 | 0 | 1 (1)
Oedema peripheral (General disorders) | 0 | 1 (2) | 2 (3)
Injection site erythema (General disorders) | 0 | 1 (3) | 1 (1)
Injection site hypersensitivity (General disorders) | 0 | 0 | 2 (3)
Fatigue (General disorders) | 0 | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 0 | 0 | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 | 0
Injection site pruritus (General disorders) | 0 | 1 (3) | 0
Injection site swelling (General disorders) | 0 | 1 (3) | 0
Injection site haematoma (General disorders) | 0 | 1 (2) | 0
Injection site induration (General disorders) | 0 | 0 | 1 (2)
Gait disturbance (General disorders) | 0 | 1 (1) | 0
Injection site pain (General disorders) | 0 | 0 | 1 (1)
Impaired healing (General disorders) | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 (1) | 0 | 1 (2)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 1 (1) | 0
Troponin T increased (Investigations) | 1 (1) | 0 | 1 (1)
Albumin urine present (Investigations) | 0 | 1 (1) | 0
Blood creatinine increased (Investigations) | 0 | 1 (1) | 0
High density lipoprotein decreased (Investigations) | 0 | 0 | 1 (1)
White blood cell count increased (Investigations) | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 (1) | 0 | 5 (14)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 (3)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)
Cardiac contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT03002974/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT03002974/SAP_001.pdf